CLINICAL TRIAL: NCT02734758
Title: Atrial Fibrillation in Ischemic Stroke: Strengthening Identification and Decisions to Anticoagulate
Brief Title: Markers of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 248994
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Atrial fibrillation stroke
- Non-atrial fibrillation Stroke

SUMMARY:
This study will evaluate whether a gene marker can improve the identification of atrial fibrillation in patients with ischemic stroke, and evaluate whether the decision to anticoagulate could be improved by a marker of atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a major cause of ischemic stroke that is critical to identify because anticoagulation provides a 66% risk reduction in recurrent stroke. However, opportunities to prevent stroke due to AF are frequently missed because AF is paroxysmal and therefore not detected at the time of stroke. In addition, even when AF is identified anticoagulation may not be initiated due to perceived contraindications.

This study will (1) evaluate whether a gene marker can improve the identification of AF in patients with ischemic stroke, and (2) evaluate decisions by health care provider and patients to anticoagulate AF, and whether this decision could be improved by a marker of AF at time of stroke. An AF Gene Score will be developed comprised of genes associated with inflammatory and thrombotic pathways related to risk of AF thromboembolism in stroke patients with AF. The AF Gene Score measured at time of stroke can stroke will permits rapid identification of stroke due to AF which may increase initiation of anticoagulation therapy. This is important in cryptogenic stroke, where prolonged monitoring leaves uncertainty regarding the association of delayed AF with initial stroke and delays anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke within 72 hours of onset
* Complete evaluation to determine cause of stroke
* Informed Consent

Exclusion Criteria:

* Active Infection
* Lymphoma / Leukemia / Blood dyscrasia
* Hemorrhagic stroke
* Immunosuppressive therapy
* Illicit drug use
* Blood transfusion +/- 1 month
* Major surgery/trauma in last 6mts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Gene expression | Post stroke through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States